CLINICAL TRIAL: NCT02318511
Title: An Investigation of ReNu™ Knee Injection: Monitoring the Response of Knee Function and Pain in Patients With Osteoarthritis
Brief Title: An Investigation of ReNu™ Knee Injection in Patients With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NuTech Medical, Inc (Industry)
Collaborators: Organogenesis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RD2014-10-04
Record Dates: First submitted 2014-12-09; First posted 2014-12-17 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- ReNu amniotic allograft (Experimental): Knee injection with ReNu. ReNu is an allograft tissue composed of particularized amniotic membrane and cell from the amniotic fluid.
  Interventions: Procedure: Knee injection; Other: ReNu amniotic allograft
- Saline (Placebo Comparator): Knee injection with saline. Injectable saline will be used as the placebo control.
  Interventions: Procedure: Knee injection; Device: placebo saline
- HA injection (Active Comparator): Knee injection with HA. HA will be used as a viscosupplementation injection consisting of cross linked HA.
  Interventions: Procedure: Knee injection; Device: Hyaluronic Acid

INTERVENTIONS:
Procedure: Knee injection — Injection into knee for the treatment of Osteoarthritis
Other: ReNu amniotic allograft
  Arms: ReNu amniotic allograft
Device: placebo saline
  Arms: Saline
Device: Hyaluronic Acid
  Arms: HA injection

SUMMARY:
This is a Prospective, Randomized study evaluating the efficacy of ReNu for the treatment of Kellgren-Lawrence grade 2 or 3 osteoarthritis. Patients will be randomized into 1 of 3 groups for injection into the effected knee: 1) ReNu - study treatment, 2) Hyaluronic Acid (HA) injection - with commonly used injection material and 3) Saline. After treatment, patients will be followed up to 12 months to evaluate improvements using common pain and function subscales.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate knee osteoarthritis determined by a combination of clinical and radiographic findings and documented by Kellgren-Lawrence radiographic classification (Grade 2 or 3)
* Grade 2 Kellgren-Lawrence radiographic changes are defined as small osteophytes, possible narrowing of joint space
* Grade 3 Kellgren-Lawrence radiographic changes are defined as moderate multiple osteophytes, definite narrowing of joints space, some sclerosis and possible deformity of bone contour.
* Patients with bilateral grade 2 or 3 Kellgren Lawrence knee osteoarthritis who have bilateral symptoms may have their more symptomatic knee injected. If equivalent symptoms are reported by the patient, then the patient will choose which knee is to be injected. The contralateral knee can be treated with local standard of care such as steroid injection, cold therapy or soft brace.
* Age 18 and older
* BMI less than 40
* 7 day average pain score of 4 or greater for the involved knee on a numeric pain scale from 1 to 10.
* Female patients must be actively practicing a contraception method, abstinence, be surgically sterilized, or be postmenopausal

Exclusion Criteria:

* Pain medication (including nonsteroidal antiinflammatory drugs, NSAIDs) less than 15 days before injection (may take acetaminophen)
* Receiving pain medication other than acetaminophen for conditions unrelated to osteoarthritis of the index knee
* Regular use of anticoagulants, such as Coumadin, dabigatran or rivaroxaban; use of antiplatelet medications are not a reason for exclusion
* History of substance abuse.
* Failure to agree NOT to take additional knee symptom modifying drugs, other than acetaminophen, during the course of the study without reporting to the study team
* Pregnancy or desire to become pregnant during study duration
* Positive pregnancy test on premenopausal subject
* Morbid obesity (defined as BMI 40 or greater)
* Symptoms of locking, intermittent block to range of motion or loose body sensation which could indicate meniscal displacement or an intraarticular loose body
* Corticosteroid injection into the index knee within 3 months
* Viscosupplement injection into the index knee within 3 months
* Knee surgery of involved index knee within 12 months
* Knee surgery contralateral knee 6 months
* Worker compensation
* Acute index knee injury (injury within 3 months)
* History of Diabetes mellitus
* History of solid organ or hematologic transplantation
* History of rheumatoid arthritis or other autoimmune disorder
* Diagnosis of a non-basal cell malignancy within the preceding 5 years
* Infection requiring antibiotic treatment within the preceding 3 months
* Current therapy with any immunosuppressive medication, including corticosteroids at a dose > 5 mg per day

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-06; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
VAS Pain Scale Change from Baseline | 3 months
VAS Pain Scale Change from Baseline | 6 months
KOOS Pain and Function Subscales Change from Baseline | 3 months
KOOS Pain and Function Subscales Change from Baseline | 6 months

SECONDARY OUTCOMES:
KOOS Pain and Function Subscales change from Baseline | 1 week, 6 weeks, 3 months, and 12 months
Other patient reported outcomes (PROs) change from Baseline | 1 week, 6 week, 3 months, 6 months, and 12 months
Radiographic (X-ray) measurement of standing joint space change from Baseline | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jack Farr, MD, Principal Investigator — OrthoIndy
Locations (12):
- United States (12):
  - American Sports Medicine Institute, Birmingham, Alabama
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Midwest Orthopedics at Rush, LLC, Chicago, Illinois
  - Orthoindy, Indianapolis, Indiana
  - Center for Clinical and Translational Science UK Chandler Medical Center, Pavilion H, Lexington, Kentucky
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Missouri Orthopaedic Institute (MOI), Columbia, Missouri
  - New Mexico Orthopaedics, Albuquerque, New Mexico
  - New York University, New York, New York
  - Hospital for Special Surgery, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Advanced Orthopedics, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No